CLINICAL TRIAL: NCT03720379
Title: Efficacy of Fluor Protector S in the Prevention of Tooth Decay in Adolescents
Brief Title: Efficacy of Fluor Protector S in the Prevention in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Warsaw (Other)
Collaborators: Ivoclar Vivadent AG (Industry); Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KB/226/2017
Record Dates: First submitted 2018-10-17; First posted 2018-10-25 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2018-10

CONDITIONS: Dental Caries; Fluor
Keywords: fluoride varnish; dental caries; ADOLESCENTS
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: We plan to include 168 subjects in this study.
  1. Dental examination Qualified for the study will receive oral and written information on the causative factors of dental caries, hygienic and dietary recommendations.
  2. Oral hygiene instruction will be provided.
  3. Caries risk assesment
  4. Application Fluor Protector S or Placebo
  Dental examination will be performed before the intervention (preliminary), after 6 months and after 12 months. Dental exams will include an interview, a physical examination , radiological examination (bite- wing x-ray images) and Diagnodent assessment.
  The applications of Fluor Protector S (intervention A) or placebo (intervention B) will be performed every three months during one year.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants,Care Providers, Investigators and Outcomes Assessor will be aware of the current subject's allocation and will be unconscious which product is fluoride varnish and which placebo. participants assigned to intervention(s) based on a protocol Patients will be distributed between Group A (Fluor Protector S) and group B (placebo) according to allocation for 2 types of intervention and blindness (codes for the type of intervention A and B will be assigned to patient numbers according to the reporting order and placed in opaque envelopes).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoride Varnish - Fluor PROTECTOR S (Active Comparator): Fluor Protector S - manufacturer: Ivoclar Vivadent Composition: ethanol, water, polymer, saccharin, mint flavor, 1.5% ammonium fluoride (7700 ppm fluoride), additional ingredients
  APPLICATION OF Fluor Protector S will be performed AT BASELINE, after 3,6 months (control 1) and after 9 and 12 months (control 2). Preliminary(AT BASELINE) and control dental exams after 12 months will include an interview and a physical examination, radiological and Diagnodent examination, a 6 months follow-up -a physical examination, Diagnodent examination and interview.
  Interventions: Device: Fluor Protector S
- PLACEBO (Placebo Comparator): - Placebo - manufacturer: Ivoclar Vivadent Composition: ethanol, water, polymer, saccharin, mint flavor.
  APPLICATION OF PLACEBO will be performed AT BASELINE, after 3,6 months (control 1) and after 9 AND 12 months (control 2). Preliminary(AT BASELINE) and control dental exams after 12 months will include an interview and a physical examination, radiological and Diagnodent examination, a 6 months follow-up -a physical examination, Diagnodent examination and interview.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Fluor Protector S — . All of the elements of a clinical trial and the varnish applications will be performed every three-month during one year: Changes in The Simplified Oral Hygiene Index (OHl-S), white spot carious lesion discovered at the initial assessment as invisible, visible and inactive, active, cavities), dmft and dmfs and their components, bite-wings and Diagnodent assessment will be scored at follow-up examinations.
  Arms: Fluoride Varnish - Fluor PROTECTOR S
Device: Placebo — All of the elements of a clinical trial and the placebo applications will be performed every three-month during one year: Changes in The Simplified Oral Hygiene Index (OHl-S), white spot carious lesion discovered at the initial assessment as invisible, visible and inactive, active, cavities), dmft and dmfs and their components, bite-wings and Diagnodent assessment will be scored at follow-up examinations.
  Arms: PLACEBO

SUMMARY:
Purpose of the study is to evaluate the effectiveness of Fluor Protector S in preventing tooth decay in adolescents and to isolate factors that reduce its effectiveness.

In this study, half of the randomly assigned participants will received fluoride varnish (Fluor Protector S) and will be considered an intervention group. The other half will undergo placebo application.

DETAILED DESCRIPTION:
Evidence from 6 systematic reviews involving 200 trials and more than 80,000 participants further supports the effectiveness of fluoride varnishes, applied professionally 2-4 times a year, for preventing dental caries. Additionally, the simultaneous use of fluoride varnishes with fluoride toothpaste appears to significantly enhance the caries-inhibiting effect compared with the use of fluoride toothpaste alone. The relative benefit of fluoride varnishes application seems to occur irrespective of baseline caries risk, baseline caries severity, background exposure to fluorides and application features such as prior prophylaxis, concentration of fluoride or frequency of application.

To determine the sample size, the results of epidemiological studies conducted in the framework of the health monitoring of the Polish population in 2015 in the group of people aged 15 years (dmf = 5.75) and in 2016 in the group of people aged 12 years (dmf = 3) 0.7 as annual growth of caries, and literature data on the effectiveness of fluoride varnish in the prevention of permanent tooth decay in the general population at 43% (a reduction of about 0.3% per year in dmf, Standard Deviation = 0.8) and was considered achievable in the case Apply Fluor Protector S at 3 months intervals in the high risk group of caries. Size of the study group with such assumptions (α = 0,05, power = 80%, mean reduction of dmf: 0,3, Standard Deviation = 0,8 ; t test for comparison of two groups) - Minimum 84 patients [70 patients+ 20% (dropped out), in both groups].

Participants will be allocated to the "test" and to the "control" group, respectively, by computer-generated randomly permuted blocks using R package in statistical software..

* The children will be examined and re-examined clinically by the same examiners.
* Statistical analyses will be performed using statistical software, the level of significance was set at 0.05. Intra-examiner reliability was assessed by kappa statistics.
* To compare average values between two independent groups U Mann-Whitney test will be used (for e.g. to compare experimental group with the control one); Wilcoxon signed-rank test will be used for paired samples (for e.g. to compare first measurement with final measurement for experimental group). Comparison of fractions will be conducted using Pearson's chi-square test of independence and Z test. The 95% confidence intervals will be calculated on the basis of normal approximation.

Purpose of the study is to evaluate the effectiveness of Fluor Protector S in preventing tooth decay in adolescents and to isolate factors that reduce its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age> 12 ≤ 19 years
* All permanent teeth (except the third molar teeth)
* Restored caries lesions
* Teeth with International Caries Detection and Assessment System II score 0, 1, or 2
* Agreement of parents / legal guardians and patients to participate in the study

Exclusion Criteria:

* Planned change of residence during the year
* Chronic illness or medication that increases the risk of tooth decay
* Orthodontic treatment
* Caries lesions

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 168 (Estimated)
Dates: Start 2018-10-19 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence and intensity of dental caries | 12 months
  The decrease of caries, which means a lower caries occurrence and intensity (lower caries index dmft/dmfs) when comparing to the placebo group.
  Diagnodent assessment scale similar at baseline and at the end of the study. The same number of teeth/surfaces with no caries in the fluoride varnish group when comparing to the placebo group, according to scale:
  0-14 No caries 15-20 Enamel caries 21-99 Dentinal caries
  In the study, bite-wing images are planned at 12 months intervals. The scale will be used to evaluate:
  E1 - carious lesion including <1/2 enamel, E2 - carious lesion including> 1/2 enamel, D1 - tooth decay in dentin, not exceeding 1/3 of dentin, D2 - caries in the middle 1/3 of dentin, D3 carious lesion > 2/3 of dentin. Codes E1 and E2 will be recorded as pre-cavity, codes ≥ D1 as cavity. Primary outcome is no signs of caries during radiological examination in fluoride varnish group when comparing to the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Olczak Kowalczyk, PROFESSOR, Study Director — Medical University of Warsaw
Locations (1):
- Dorota Olczak-Kowalczyk, Warsaw, Warsaw, 18 Miodowa Saint, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lenzi TL, Montagner AF, Soares FZ, de Oliveira Rocha R. Are topical fluorides effective for treating incipient carious lesions?: A systematic review and meta-analysis. J Am Dent Assoc. 2016 Feb;147(2):84-91.e1. doi: 10.1016/j.adaj.2015.06.018. Epub 2015 Nov 6. PMID 26562737
- [Background] Bansal A, Ingle NA, Kaur N, Ingle E. Recent advancements in fluoride: A systematic review. J Int Soc Prev Community Dent. 2015 Sep-Oct;5(5):341-6. doi: 10.4103/2231-0762.165927. PMID 26539383
- [Background] Weyant RJ, Tracy SL, Anselmo TT, Beltran-Aguilar ED, Donly KJ, Frese WA, Hujoel PP, Iafolla T, Kohn W, Kumar J, Levy SM, Tinanoff N, Wright JT, Zero D, Aravamudhan K, Frantsve-Hawley J, Meyer DM; American Dental Association Council on Scientific Affairs Expert Panel on Topical Fluoride Caries Preventive Agents. Topical fluoride for caries prevention: executive summary of the updated clinical recommendations and supporting systematic review. J Am Dent Assoc. 2013 Nov;144(11):1279-91. doi: 10.14219/jada.archive.2013.0057. PMID 24177407
- [Background] Richards D. Substantial reduction in caries from regular fluoride varnish application. Evid Based Dent. 2013 Sep;14(3):72-3. doi: 10.1038/sj.ebd.6400947. PMID 24071672
- [Background] Gao SS, Zhang S, Mei ML, Lo EC, Chu CH. Caries remineralisation and arresting effect in children by professionally applied fluoride treatment - a systematic review. BMC Oral Health. 2016 Feb 1;16:12. doi: 10.1186/s12903-016-0171-6. PMID 26831727
- [Background] Marinho VC, Worthington HV, Walsh T, Clarkson JE. Fluoride varnishes for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2013 Jul 11;2013(7):CD002279. doi: 10.1002/14651858.CD002279.pub2. PMID 23846772